CLINICAL TRIAL: NCT03863067
Title: Assessment Of Clinical Effectiveness, Security And Correlation With Radiological Changes In Patients With Lumbar Stenosis Treated With Epiduroscopy
Brief Title: Clinical Effectiveness, Security And Radiological Changes In Epiduroscopy For Lumbar Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIC131-18
Record Dates: First submitted 2019-01-21; First posted 2019-03-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Spinal Stenosis, Lumbar Region, With Neurogenic Claudication
Keywords: Lumbosacral epiduroscopy; spinal stenosis; magnetic resonance imaging; intraoperative neurophysiological monitoring; neurogenic claudication
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lumbar spinal stenosis patients (Experimental): Epiduroscopy in patients with lumbar spinal stenosis
  Interventions: Procedure: Epiduroscopy

INTERVENTIONS:
Procedure: Epiduroscopy — Using epiduroscopy to treat the ligamentum flavum hypertrophy with Resaflex ,an instrument with Quantum Molecular Resonance for tissue coablation.
  Other Names: Spinal endoscopy

SUMMARY:
It will be done a prospective Study involving 38 patients with lumbar stenosis. A magnetic resonance (MR) imaging study and a electromyographic study will be done previously and 3 months after the epiduroscopy to confirm radiologic or neurophysiological changes.

During the technic it will be used different instruments, an endoscope developed for its use in the epidural space (Resascope), a Fogarty balloon (Resaloon) to dilate the space near the epidural recess where it will be try to decrease the ligamentum flavum using the Resaflex, an instrument with Quantum Molecular Resonance for tissue coablation, in order to get less symptomatic lumbar stenosis.

The investigators will compare qualitative and quantitative variables at baseline and 1, 3, 6, ant 12 months after the epiduroscopy.

DETAILED DESCRIPTION:
The investigators perform the Interventional Endoscopic Spinal Surgical (IESS) ,with the different instruments mentioned above. The Resaflex wich use Quantum Molecular Resonance, through combination of different frequencies in the range of the radio-frequency, emit quantum in resonance and produce lesion and coagulation; The objective is to reach the ligamentum flavum doing lesions to diminish the stenosis caused by hypertrophic ligamentum over all in the recess area near the radicular nerve.

To increase the security of the procedure the investigators introduce for the first time , neurophysiological monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication for epiduroscopy in the usual clinical practice
* Neurogenic claudication
* Lumbar pain for more than 6 months
* Numerical rating scale >6
* No response with medical treatment
* No response with other interventional treatment: epidurolysis

Exclusion Criteria:

* Psychiatric disorders
* Opioid addiction
* Acute organic disease
* Severe chronic organic disease
* Vasculo-cerebral disease
* Coagulation alterations
* Ofthalmologic disease
* Allergic
* Infections
* Impossibility to understand the procedure

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Quantitative measurements in lumbar magnetic resonance imaging | Baseline
  Measure in mm of ligamentum flavum at the level with major stenosis at the medium area of the ligamentum and in the recess
Quantitative measurements in lumbar magnetic resonance imaging | Three months after the technic
  Measure in mm of ligamentum flavum at the level with major stenosis at the medium area of the ligamentum and in the recess
Qualitative changes in lumbar magnetic resonance imaging | Baseline
  Schizas classification( A:no stenosis, B: moderate; C:severe) at the level where there are major stenosis
Qualitative changes in lumbar magnetic resonance imaging | three months after the technic
  Schizas classification( A:no stenosis, B: moderate; C:severe) at the level where there are major stenosis
Numerical rating scale | Baseline
  Pain from 0 (no pain) to 10 (worst pain imaginable)
Numerical rating scale | 1 month after the technic
  Pain from 0 (no pain) to 10 (worst pain imaginable)
Numerical rating scale | 3 months after the technic
  Pain from 0 (no pain) to 10 (worst pain imaginable)
Numerical rating scale | 6 months after the technic
  Pain from 0 (no pain) to 10 (worst pain imaginable)
Numerical rating scale | 12 months after the technic
  Pain from 0 (no pain) to 10 (worst pain imaginable)
Likert Scale to record the percentage of improvement | baseline
  Percentage of improvement: 1 (>75% worst) 2 >50% worst; 3 (>25% worst); 4 (no changes); 5 ( 25% better); 6 (50% better); 7 (75% better)
Likert Scale to record the percentage of improvement | 1 month after the technic
  Percentage of improvement: 1 (>75% worst) 2 >50% worst; 3 (>25% worst); 4 (no changes); 5 ( 25% better); 6 (50% better); 7 (75% better)
Likert Scale to record the percentage of improvement | 3 months after the technic
  Percentage of improvement: 1 (>75% worst) 2 >50% worst; 3 (>25% worst); 4 (no changes); 5 ( 25% better); 6 (50% better); 7 (75% better)
Likert Scale to record the percentage of improvement | 6 months after the technic
  Percentage of improvement: 1 (>75% worst) 2 >50% worst; 3 (>25% worst); 4 (no changes); 5 ( 25% better); 6 (50% better); 7 (75% better)
Likert Scale to record the percentage of improvement | 12 months after the technic
  Percentage of improvement: 1 (>75% worst) 2 >50% worst; 3 (>25% worst); 4 (no changes); 5 ( 25% better); 6 (50% better); 7 (75% better)
EuroQualityofLife visual analogue scale (EQ VAS) | Baseline
  The EQ visual analogue scale (EQ VAS). VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints wich comes from 0 to 100 are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). This can be used as a quantitative measure of health outcome. The higher values indicates a better outcome.
EuroQualityofLife Five-Dimensions Five-Levels Questionnaire(EQ-5D-5L) | Baseline
  The 5-level EQ-5D version (EQ-5D-5L) consists of:
  1- The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
EuroQualityofLife visual analogue scale (EQ VAS) | 1 month after
  The EQ visual analogue scale (EQ VAS). VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints wich comes from 0 to 100 are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). This can be used as a quantitative measure of health outcome. The higher values indicates a better outcome.
EuroQualityofLife Five-Dimensions Five-Levels Questionnaire(EQ-5D-5L) | 1 month after
  The 5-level EQ-5D version (EQ-5D-5L) consists of:
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
EuroQualityofLife visual analogue scale (EQ VAS) | 3 months after
  The EQ visual analogue scale (EQ VAS). VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints wich comes from 0 to 100 are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). This can be used as a quantitative measure of health outcome. The higher values indicates a better outcome.
EuroQualityofLife Five-Dimensions Five-Levels Questionnaire(EQ-5D-5L) | 3 months after
  The 5-level EQ-5D version (EQ-5D-5L) consists of:
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
EuroQualityofLife visual analogue scale (EQ VAS) | 6 months after
  The EQ visual analogue scale (EQ VAS). VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints wich comes from 0 to 100 are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). This can be used as a quantitative measure of health outcome. The higher values indicates a better outcome.
EuroQualityofLife Five-Dimensions Five-Levels Questionnaire(EQ-5D-5L) | 6 months after
  The 5-level EQ-5D version (EQ-5D-5L) consists of:
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
EuroQualityofLife visual analogue scale (EQ VAS) | 12 months after
  The EQ visual analogue scale (EQ VAS). VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints wich comes from 0 to 100 are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). This can be used as a quantitative measure of health outcome. The higher values indicates a better outcome.
EuroQualityofLife Five-Dimensions Five-Levels Questionnaire(EQ-5D-5L) | 12 months after
  The 5-level EQ-5D version (EQ-5D-5L) consists of:
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Oswestry Disability Index (ODI) | Baseline
  Low back pain disability questionnaire: is a validated, 10-point patient-reported outcome questionnaire. It is considered the 'gold standard' for measuring disability and quality of life (QoL) impairment for adults with low back pain (LBP).The 10 factors which constitute the ODI criteria for assessing patients' functional impairment are pain intensity, ease of personal care, lifting, working, sitting, stand-ing, sleeping, sex life, social life and travelling. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity: 0-20, minimal disability; 21-40, moderate disability; 41-60, severe disability; 61-80, crippling back pain; 81-100, these patients are either bed-bound or have an exaggeration of their symptoms. In order for the results to be deemed clinically significant, a change in the patient's score of 10% or more is required
Oswestry Disability Index (ODI) | 1 month after
  Low back pain disability questionnaire: is a validated, 10-point patient-reported outcome questionnaire. It is considered the 'gold standard' for measuring disability and quality of life (QoL) impairment for adults with low back pain (LBP).The 10 factors which constitute the ODI criteria for assessing patients' functional impairment are pain intensity, ease of personal care, lifting, working, sitting, stand-ing, sleeping, sex life, social life and travelling. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity: 0-20, minimal disability; 21-40, moderate disability; 41-60, severe disability; 61-80, crippling back pain; 81-100, these patients are either bed-bound or have an exaggeration of their symptoms. In order for the results to be deemed clinically significant, a change in the patient's score of 10% or more is required
Oswestry Disability Index (ODI) | 3 months after
  Low back pain disability questionnaire: is a validated, 10-point patient-reported outcome questionnaire. It is considered the 'gold standard' for measuring disability and quality of life (QoL) impairment for adults with low back pain (LBP).The 10 factors which constitute the ODI criteria for assessing patients' functional impairment are pain intensity, ease of personal care, lifting, working, sitting, stand-ing, sleeping, sex life, social life and travelling. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity: 0-20, minimal disability; 21-40, moderate disability; 41-60, severe disability; 61-80, crippling back pain; 81-100, these patients are either bed-bound or have an exaggeration of their symptoms. In order for the results to be deemed clinically significant, a change in the patient's score of 10% or more is required
Oswestry Disability Index (ODI) | 6 months after
  Low back pain disability questionnaire: is a validated, 10-point patient-reported outcome questionnaire. It is considered the 'gold standard' for measuring disability and quality of life (QoL) impairment for adults with low back pain (LBP).The 10 factors which constitute the ODI criteria for assessing patients' functional impairment are pain intensity, ease of personal care, lifting, working, sitting, stand-ing, sleeping, sex life, social life and travelling. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity: 0-20, minimal disability; 21-40, moderate disability; 41-60, severe disability; 61-80, crippling back pain; 81-100, these patients are either bed-bound or have an exaggeration of their symptoms. In order for the results to be deemed clinically significant, a change in the patient's score of 10% or more is required
Oswestry Disability Index (ODI) | 12 months after
  Low back pain disability questionnaire: is a validated, 10-point patient-reported outcome questionnaire. It is considered the 'gold standard' for measuring disability and quality of life (QoL) impairment for adults with low back pain (LBP).The 10 factors which constitute the ODI criteria for assessing patients' functional impairment are pain intensity, ease of personal care, lifting, working, sitting, stand-ing, sleeping, sex life, social life and travelling. Each of the 10 questions is scored from 0 to 5, giving a maximum score of 50. The total score is then converted into a percentage by multiplying it by 2. Scores are stratified into severity: 0-20, minimal disability; 21-40, moderate disability; 41-60, severe disability; 61-80, crippling back pain; 81-100, these patients are either bed-bound or have an exaggeration of their symptoms. In order for the results to be deemed clinically significant, a change in the patient's score of 10% or more is required
Zurich questionnaire | Baseline
  Claudication test:The scale relates to symptoms over the past month. There are 12 questions for all patients, and a further 6 questions to measure treatment outcome (for those who have had treatment).
  The The Zurich Claudication Questionnaire consists of three subscales:
  1. Symptom severity scale (questions I-VII) [further subdivided into pain domain (questions I-IV) and a neuroischemic domain (questions V-VII)]: Possible range of the score is 1 to 5.
  2. Physical function scale (questions VIII-XII): Possible range of scores is 1 to 4.
  3. Patient's satisfaction with treatment scale (questions XIII-XVIII): the range of the scale is 1 to 4.
Zurich questionnaire | 1 month after
  Claudication test:The scale relates to symptoms over the past month. There are 12 questions for all patients, and a further 6 questions to measure treatment outcome (for those who have had treatment).
  The The Zurich Claudication Questionnaire consists of three subscales:
  1. Symptom severity scale (questions I-VII) [further subdivided into pain domain (questions I-IV) and a neuroischemic domain (questions V-VII)]: Possible range of the score is 1 to 5.
  2. Physical function scale (questions VIII-XII): Possible range of scores is 1 to 4.
  3. Patient's satisfaction with treatment scale (questions XIII-XVIII): the range of the scale is 1 to 4.
Zurich questionnaire | 3 months after
  Claudication test:The scale relates to symptoms over the past month. There are 12 questions for all patients, and a further 6 questions to measure treatment outcome (for those who have had treatment).
  The The Zurich Claudication Questionnaire consists of three subscales:
  1. Symptom severity scale (questions I-VII) [further subdivided into pain domain (questions I-IV) and a neuroischemic domain (questions V-VII)]: Possible range of the score is 1 to 5.
  2. Physical function scale (questions VIII-XII): Possible range of scores is 1 to 4.
  3. Patient's satisfaction with treatment scale (questions XIII-XVIII): the range of the scale is 1 to 4.
Zurich questionnaire | 6 months after
  Claudication test:The scale relates to symptoms over the past month. There are 12 questions for all patients, and a further 6 questions to measure treatment outcome (for those who have had treatment).
  The The Zurich Claudication Questionnaire consists of three subscales:
  1. Symptom severity scale (questions I-VII) [further subdivided into pain domain (questions I-IV) and a neuroischemic domain (questions V-VII)]: Possible range of the score is 1 to 5.
  2. Physical function scale (questions VIII-XII): Possible range of scores is 1 to 4.
  3. Patient's satisfaction with treatment scale (questions XIII-XVIII): the range of the scale is 1 to 4.
Zurich questionnaire | 12 months after
  Claudication test:The scale relates to symptoms over the past month. There are 12 questions for all patients, and a further 6 questions to measure treatment outcome (for those who have had treatment).
  The The Zurich Claudication Questionnaire consists of three subscales:
  1. Symptom severity scale (questions I-VII) [further subdivided into pain domain (questions I-IV) and a neuroischemic domain (questions V-VII)]: Possible range of the score is 1 to 5.
  2. Physical function scale (questions VIII-XII): Possible range of scores is 1 to 4.
  3. Patient's satisfaction with treatment scale (questions XIII-XVIII): the range of the scale is 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: DAVID ABEJON, MD, PHD, Study Director — HOSPITAL QUIRONSALUD MADRID
Locations (1):
- Unidad de Investigación Clínica Secretaría Técnica CEImFJD Hospital Universitario Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manchikanti L, Saini B, Singh V. Spinal endoscopy and lysis of epidural adhesions in the management of chronic low back pain. Pain Physician. 2001 Jul;4(3):240-65. PMID 16900252
- [Background] Raffaeli W, Righetti D, Andruccioli J, Sarti D. Periduroscopy: general review of clinical features and development of operative models. Acta Neurochir Suppl. 2011;108:55-65. doi: 10.1007/978-3-211-99370-5_10. PMID 21107939
- [Background] Deyo RA. Treatment of lumbar spinal stenosis: a balancing act. Spine J. 2010 Jul;10(7):625-7. doi: 10.1016/j.spinee.2010.05.006. PMID 20620984
- [Background] Kalichman L, Cole R, Kim DH, Li L, Suri P, Guermazi A, Hunter DJ. Spinal stenosis prevalence and association with symptoms: the Framingham Study. Spine J. 2009 Jul;9(7):545-50. doi: 10.1016/j.spinee.2009.03.005. Epub 2009 Apr 23. PMID 19398386
- [Background] Chad DA. Lumbar spinal stenosis. Neurol Clin. 2007 May;25(2):407-18. doi: 10.1016/j.ncl.2007.01.003. PMID 17445736
- [Background] Raffaeli W, Righetti D. Surgical radio-frequency epiduroscopy technique (R-ResAblator) and FBSS treatment: preliminary evaluations. Acta Neurochir Suppl. 2005;92:121-5. doi: 10.1007/3-211-27458-8_26. PMID 15830982
- [Derived] Monzon EM, Rios A, Carrascoso J, Moreno P, Abejon D. Epiduroscopy in spinal stenosis. Description of the procedure and safety measures to reduce complications. Pain Manag. 2025 Nov;15(11):827-834. doi: 10.1080/17581869.2025.2552636. Epub 2025 Sep 8. PMID 40920478